CLINICAL TRIAL: NCT04559321
Title: Comparison of the 100 W Holmium Laser Lithotripsy Rate Versus LithoClast Trilogy EMS in Percutaneous Mini-nephrolithotomy for Patients With Kidney Stones GUY's 1 and 2: Randomized Clinical Trial
Brief Title: Holmium Vs Trilogy Kidney Stones GUY's 1-2
Acronym: TriHolmium
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Regional de Alta Especialidad del Bajio (Other)
Collaborators: Braulio Omar Manzo Pérez (Unknown); Edson Dazaeb Flores Hernández (Unknown); Pompeyo Stalin Alarcón Vigil (Unknown)
Responsible Party: Principal Investigator, Edgard Lozada, Master in clinical research, Hospital Regional de Alta Especialidad del Bajio
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CI-HRAEB-056-2020
Record Dates: First submitted 2020-09-04; First posted 2020-09-22 (Actual); Last update posted 2020-09-22 (Actual); Status verified 2020-09

CONDITIONS: Kidney Stone; Kidney Calculi; Kidney Diseases
Keywords: Kidney Calculi
MeSH Terms: conditions — Kidney Calculi; Kidney Diseases

STUDY DESIGN:
Intervention Model Description: 116 cases will be subjected to a simple randomization with a table of random numbers, 58 patients will undergo a percutaneous mini nephrolithotomy and lithotripsy with LithoClast Trilogy EMS; and the remaining 58 will undergo 100W Holmium laser lithotripsy.
Who Masked: Participant, Outcomes Assessor
Masking Description: Double-blind. Patient and doctor who performs the statistical analysis will not know which group each patient belongs to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Holmium laser (Active Comparator): General anesthesia, Valdivia-Galdakao position, cystoscopy will be performed, ascending pyelography will be performed. A systematic nephroscopy will be performed and once the calculation will proceed to its fragmentation with 100 W Holmium laser.
  Interventions: Procedure: Fragmentation of calculi with 100 W Holmium laser or LithoClast Trilogy EMS and 1.5 mm x 440 mm probe, according to randomization.
- Trilogy (Experimental): General anesthesia, Valdivia-Galdakao position, cystoscopy will be performed, ascending pyelography will be performed. A systematic nephroscopy will be performed and once the calculation will proceed to its fragmentation with LithoClast Trilogy EMS and 1.5 mm x 440 mm probe
  Interventions: Procedure: Fragmentation of calculi with 100 W Holmium laser or LithoClast Trilogy EMS and 1.5 mm x 440 mm probe, according to randomization.

INTERVENTIONS:
Procedure: Fragmentation of calculi with 100 W Holmium laser or LithoClast Trilogy EMS and 1.5 mm x 440 mm probe, according to randomization. — General anesthesia, Valdivia-Galdakao position, cystoscopy and ascending pyelography will be performed. A systematic nephroscopy will be performed and once the calculation will proceed to its fragmentation with 100 W Holmium laser or LithoClast Trilogy EMS and 1.5 mm x 440 mm probe, according to randomization
  Other Names: Trilogy Vs Laser Holmium

SUMMARY:
The desire to reduce complications related to percutaneous access and morbidity related to tract size has led researchers to evaluate PCNL using smaller-caliber instruments. In this context, mini-PCNL has emerged. Its efficacy and safety have been demonstrated at the cost of a lower stone-free rate.

The effectiveness of existing Ho: YAG lasers is limited by the need for manual removal of stone fragments and mobilization of them due to the lack of a simultaneous aspiration system. Consequently, this has been associated with long surgical times to achieve stone-free status. This requires multiple insertions and extractions of the nephroscope to facilitate the recovery of all fragments. This repeated step can cause the safety rails to be inadvertently removed or the sheaths to be disinserted. Sometimes compromising surgical results.

Faced with this situation, the search for better and more efficient energy sources still continues. With this, modern lithotripters have emerged that combine energy sources and work more efficiently than any of them independently and, consequently, improve stone removal. Cyberwand ™ (Olympus, Tokyo, Japan), Swiss Lithoclast® Master / Select (EMS SA, Switzerland / Boston Scientific, Marlborough, MA, USA) and Shockpulse-SE ™ (Olympus, Tokyo, Japan) are some examples; although they have their own set of advantages, none have proven to be superior to any other.

As previously discussed, ballistic-ultrasonic lithotripsy combines ultrasonic and ballistic energy together with a suction system with encouraging results in terms of a shorter lithotripsy time and the respective economic impact of fewer surgical events and less operating time required for the stone removal.

Therefore, it is convenient to make a comparison between the results of lithotripsy with Ho: YAG laser energy and lithotripsy with LithoClast Trilogy EMS; and thereby determine which is the most effective method in the resolution of kidney stones through a miniaturized percutaneous tract.

DETAILED DESCRIPTION:
Background The tools used for fragmentation and stone extraction have been improving over time. Commonly available lithotripsy power sources are classified as ultrasonic, kinetic, electrohydraulic, or combination, however, laser is the most widely used lithotripsy device in mini-PCNL as it is a small diameter power source.

Laser lithotripsy The holmium laser has been very effective in the fragmentation of stones of variable hardness and very safe due to its low depth of penetration (0.5 mm).

One of the advantages of the Ho: YAG laser is that it offers relatively quick lithotripsy while minimizing tissue trauma. Furthermore, it is effective against all stone compositions, including cystine and calcium oxalate monohydrate, where ultrasonic lithotripsy may have difficulties.

The removal of smaller fragments is possible using a vacuum effect where the fragments are moved from a high pressure zone in the pyelocaliceal system to a lower pressure zone in the sheath. If there are too many fragments, this requires multiple insertions and extractions of the nephroscope to facilitate the recovery of all of them. This repeated step can cause inadvertent movements that affect the results.

Combined ballistic-ultrasonic lithotripsy LithoClast Trilogy EMS is the newest model of percutaneous lithotripsy technology that provides electromagnetic and ultrasonic ballistic energy, as well as suction capacity under the control of the surgeon through a single pedal. Laboratory studies have suggested that combined ballistic-ultrasonic lithotripsy offers faster stone clearance than other combined and ultrasonic devices. In an in vitro comparison, LithoClast Trilogy EMS had the fastest average removal time of 23.79 seconds. This was followed by ShockPulse (46.04 seconds), Select-US (54.86 seconds), and Select-USP (102.48 seconds).

In a multi-institutional study, LithoClast Trilogy EMS was evaluated, the experience of surgeons with this device was perceived as highly satisfactory, with an excellent safety and durability profile. The average stone removal rate was 68.9 mm2 / minute. High tissue safety and an optimized aspiration configuration were reported in a prospective clinical trial. In this study, the mean stone volume clearance ratios were 370.5 ± 171 mm3 / min and 590.7 ± 250 mm3 / min for mini-PCNL and PCNL, respectively.

LithoClast Trilogy EMS has a single probe design and connects to the handpiece and oscillates with a piezoelectric ultrasonic generator at a rate of 24 kHz. At the same time, an electromagnetic generator produces ballistic motion of the entire probe at an adjustable speed of up to 12 Hz. As with other ultrasound-based devices, suction is available through the hollow probe, with the foot pedal controlling the aspiration and activation of lithotripsy. The strength of the ultrasonic vibration, the aspiration and the ballistic energy discharge frequency are adjustable through a touch screen on the generator. Various probe sizes are available (3.3 F, 4.5 F, 5.7 F, 10.2 F, and 11.7 F catheter).

JUSTIFICATION The desire to reduce complications related to percutaneous access and morbidity related to tract size has led researchers to evaluate PCNL using smaller-caliber instruments. In this context, mini-PCNL has emerged. Its efficacy and safety have been demonstrated at the cost of a lower stone-free rate.

The effectiveness of existing Ho: YAG lasers is limited by the need for manual removal of stone fragments and mobilization of them due to the lack of a simultaneous aspiration system. Consequently, this has been associated with long surgical times to achieve stone-free status. This requires multiple insertions and extractions of the nephroscope to facilitate the recovery of all fragments. This repeated step can cause the safety rails to be inadvertently removed or the sheaths to be disinserted. Sometimes compromising surgical results.

Faced with this situation, the search for better and more efficient energy sources still continues. With this, modern lithotripters have emerged that combine energy sources and work more efficiently than any of them independently and, consequently, improve stone removal. Cyberwand ™ (Olympus, Tokyo, Japan), Swiss Lithoclast® Master / Select (EMS SA, Switzerland / Boston Scientific, Marlborough, MA, USA) and Shockpulse-SE ™ (Olympus, Tokyo, Japan) are some examples; although they have their own set of advantages, none have proven to be superior to any other.

As previously discussed, ballistic-ultrasonic lithotripsy combines ultrasonic and ballistic energy together with a suction system with encouraging results in terms of a shorter lithotripsy time and the respective economic impact of fewer surgical events and less operating time required for the stone removal.

Therefore, it is convenient to make a comparison between the results of lithotripsy with Ho: YAG laser energy and lithotripsy with LithoClast Trilogy EMS; and thereby determine which is the most effective method in the resolution of kidney stones through a miniaturized percutaneous tract.

PROBLEM STATEMENT What is the difference of the lithotripsy rate with LithoClast Trilogy EMS compared to 100 W Holmium laser for patients with kidney stones GUY's 1 and 2 in percutaneous mini nephrolithotomy?

HYPOTHESIS H0: Lithotripsy performed with LithoClast Trilogy EMS in patients with GUY's 1 and 2 kidney stones undergoing percutaneous mini nephrolithotomy has a higher lithotripsy rate than that performed with a 100W Holmium laser.

Hi: Lithotripsy performed with LithoClast Trilogy EMS in patients with GUY's 1 and 2 kidney stones undergoing percutaneous mini nephrolithotomy has a lower lithotripsy rate than that performed with a 100W Holmium laser.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients older than 18 years
* Diagnosis of GUY´s kidney stones 1 and 2 who will undergo a percutaneous mini nephrolithotomy
* Preoperative serum hemoglobin> 10 g / dl
* Preoperative serum creatinine <1.5 mg / dl.
* Surgical risk I-III according to "American Society of Anesthesiologists".
* Previous negative urine culture.
* With postoperative follow-up with computed tomography at three months.
* Patients who are not participating in another project related to the treatment of lithiasis -Who have signed an informed consent where they agree to be part of the study.

Exclusion Criteria:

* Patients with a history of coagulopathies.
* Patients with anatomical abnormalities of the urinary tract.
* Pregnant patients.
* Patients with kidney stones GUY´s 3 and 4.
* Patients who do not wish to participate in the clinical trial.
* Patient who due to their physical and / or mental state are not able to sign the informed consent.

Elimination criteria. Patients who have lost follow-up in the first three months after treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-09-30 (Estimated); Primary Completion 2021-09-02 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Stone clearance | 10 minutes
  defined as the kidney stone surface area in square millimeters measured by pre-operative computed tomography scan divided by the time to remove the targeted stone burden in minutes

SECONDARY OUTCOMES:
Complications during surgery | 3 months
  All complications measured by the Clavien Classification of Surgical Complications during surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Edgard Efren Dr Lozada Hernandez, Master, Study Director — Hospital Regional de Alta Especialidad
Locations (1):
- Hospital Regional de Alta Especilidad del bajio, León, Guanajuato, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Via email, any researcher may request the database.
Supporting Information: Study Protocol, ICF
Time Frame: From the beginning of the study to its end
Access Criteria: Via email, any researcher may request the documents.

REFERENCES:
- [Result] Scotland KB, Kroczak T, Pace KT, Chew BH. Stone technology: intracorporeal lithotripters. World J Urol. 2017 Sep;35(9):1347-1351. doi: 10.1007/s00345-017-2057-x. Epub 2017 Jun 12. PMID 28608192
- [Result] Vassar GJ, Chan KF, Teichman JM, Glickman RD, Weintraub ST, Pfefer TJ, Welch AJ. Holmium: YAG lithotripsy: photothermal mechanism. J Endourol. 1999 Apr;13(3):181-90. doi: 10.1089/end.1999.13.181. PMID 10360498
- [Result] Okhunov Z, del Junco M, Yoon R, Labadie K, Lusch A, Ordon M. In vitro evaluation of LithAssist: a novel combined holmium laser and suction device. J Endourol. 2014 Aug;28(8):980-4. doi: 10.1089/end.2014.0111. Epub 2014 May 8. PMID 24707884
- [Result] Dauw CA, Borofsky MS, York N, Lingeman JE. A Usability Comparison of Laser Suction Handpieces for Percutaneous Nephrolithotomy. J Endourol. 2016 Nov;30(11):1165-1168. doi: 10.1089/end.2016.0203. PMID 27758119
- [Result] Carlos EC, Wollin DA, Winship BB, Jiang R, Radvak D, Chew BH, Gustafson MR, Simmons WN, Zhong P, Preminger GM, Lipkin ME. In Vitro Comparison of a Novel Single Probe Dual-Energy Lithotripter to Current Devices. J Endourol. 2018 Jun;32(6):534-540. doi: 10.1089/end.2018.0143. Epub 2018 May 11. PMID 29649900
- [Result] Nottingham CU, Large T, Cobb K, Sur RL, Canvasser NE, Stoughton CL, Krambeck AE. Initial Clinical Experience with Swiss LithoClast Trilogy During Percutaneous Nephrolithotomy. J Endourol. 2020 Feb;34(2):151-155. doi: 10.1089/end.2019.0561. Epub 2019 Nov 12. PMID 31588790
- [Result] Sabnis RB, Balaji SS, Sonawane PL, Sharma R, Vijayakumar M, Singh AG, Ganpule AP, Desai MR. EMS Lithoclast Trilogy: an effective single-probe dual-energy lithotripter for mini and standard PCNL. World J Urol. 2020 Apr;38(4):1043-1050. doi: 10.1007/s00345-019-02843-2. Epub 2019 Jun 8. PMID 31177306
- [Result] Wollin DA, Lipkin ME. Emerging Technologies in Ultrasonic and Pneumatic Lithotripsy. Urol Clin North Am. 2019 May;46(2):207-213. doi: 10.1016/j.ucl.2018.12.006. PMID 30961854
- [Derived] Manzo BO, Lozada Hernandez EE, Casale AR, Jimenez CJ, Gomez YR, Galvan JP, Alarcon P, Flores E, Mendez DM, Sanchez HM. Trilogy vs 100 W Ho: YAG Laser for Lithotripsy in Mini-Percutaneous Nephrolithotomy: Superior Stone-Free Rates in a Randomized Controlled Trial. Urology. 2025 Aug;202:18-24. doi: 10.1016/j.urology.2025.04.005. Epub 2025 Apr 8. PMID 40210001

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-09-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT04559321/Prot_SAP_ICF_000.pdf